CLINICAL TRIAL: NCT03460730
Title: Dynamics of the Immune Response in Children to the 23-valent Pneumococcal Capsular Polysaccharide Vaccine (Pneumovax)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Principal Investigator, Anthony Scott, Prof Anthony Scott, KEMRI-Wellcome Trust Collaborative Research Program
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEMRI_CT_2018\0022; SSC 613 (Other: KEMRI)
Record Dates: First submitted 2018-02-20; First posted 2018-03-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Pneumonia, Pneumococcal
Keywords: Invasive Pneumococcal Disease
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunised children (Experimental): Single 0.5 ml sub-cutaneous dose of 23-valent pneumococcal polysaccharide vaccine (Pneumovax)
  Interventions: Biological: Pneumovax

INTERVENTIONS:
Biological: Pneumovax — 23-valent pneumococcal polysaccharide vaccine

SUMMARY:
To explore a further dimension of susceptibility to disease, the investigators tested the hypothesis that natural variation exists in the rapidity of IgG responses following exposure to pneumococcal polysaccharides, and that these differences are sufficiently great to affect susceptibility to and outcome of IPD. The study recruited children aged 24-36 months, who had recovered from IPD, and age-matched healthy controls and vaccinated them with 1 dose of the 23-valent PPV to mimic natural exposure. The investigators collected serum samples after vaccination and analysed the dynamics of anti-polysaccharide antibody responses to several capsular antigens.

DETAILED DESCRIPTION:
The details are as described below:

1. Study site Kilifi District Hospital.
2. Study population and sampling Cases and controls from the Kilifi Birth Cohort who are alive at the end of the cohort observation (at the age of 24 months) and remain resident in Kilifi District will be vaccinated with a single 0.5 ml sub-cutaneous dose of 23 valent pneumococcal polysaccharide vaccine (Pneumovax 23) to compare the dynamics of the anti-capsular antibody response to 5 capsular antigens chosen to represent different immunological profiles of the pneumococcal capsular polysaccharides (1, 6B, 14, 19F, 23F).
3. Recruitment Potential study subjects will be identified and their mothers will be approached, informed about the study, including the necessity to undergo HIV testing, and invited to take part. A fieldworker will explain the rationale and procedures for the study and will give the mother an information sheet/consent form to take away. The mother will also be given an appointment slip and a fare to return to the hospital on the appointment date. Appointments will be at ward 1. When the mother returns the fieldworker will go through the consent form again and will ask the mother to sign. The mother will be counselled and her child will be HIV tested. If the participant is positive the child will be referred to the Kilifi Family Clinic. If the participant is negative, the child will receive the single dose of Pneumovax (23 valent polysaccharide vaccine). The mother will be given a schedule of 2 further appointments for blood tests and at each visit the fare to and from the hospital will be provided by KEMRI. Study subjects who have been vaccinated and subsequently do not attend will be visited by FW on a motorcycle to invite them to keep their appointments the very next day. Information will be collected concerning age, sex and environmental exposures such as: number of elder and younger sibling in the house, cooking smoke exposure, passive cigarette smoking, recent admission to hospital.

   Definition of cases:

   Cases of IPD, ARI or radiographic pneumonia and meningitis will be defined as episodes of illness, requiring admission to hospital, that occur to cohort members between birth and the age of 23 months that also meet at least one of the following syndrome definitions: INVASIVE PNEUMOCOCCAL DISEASE is defined by a positive result on EITHER of the following criteria: (i) culture of S. pneumoniae from any normally sterile site including blood, CSF, lung, synovial fluid but excluding middle ear fluid and external eye swabs. OR (ii) Two-fold rise in anti-PsaA antibody concentration measured by ELISA in two serum samples obtained at least 5 days apart 21 AND presence in urine of pneumococcal capsular polysaccharide detected by latex agglutination assay 46. ARI is defined by an acute (<2 weeks) history of cough or difficulty in breathing accompanied by a raised respiratory rate (≥50/min in a child <12 months, ≥40/min in a child 12-23 months). ARI is severe if there is, in addition, chest indrawing, and very severe if there is, in addition, central cyanosis and prostration or inability to drink 47.

   RADIOGRAPHIC PNEUMONIA is defined as ARI accompanied by radiographic consolidation. All radiographs will be rated both by study physicians and by a consultant radiologist. "Radiographic consolidation" will only be considered to be present if documented by both observers.

   MENINGITIS: Meningitis is being defined to target the use of additional diagnostic tests for IPD. A definition is required which is sensitive but not necessarily highly specific for pneumococcal meningitis. Any child that is transferred to the KEMRI high dependency unit with a clinical diagnosis of "Meningitis", any child started on the standard meningitis antibiotic regime, or any child with an elevated CSF leucocyte count or CSF/plasma glucose ratio of <0.5 will be considered as a case of meningitis for the purposes of this study.

   A single episode of illness may satisfy one, two, three or all case definitions. The definition of IPD is for use in the case-control study. The other definitions are for use in the study of incidence and aetiology of severe ARI and radiographic pneumonia and to guide the flow of investigations of patients with suspected IPD.
4. Laboratory Methods ANTI-CAPSULAR IGG ELISA. The method of Quataert et al. will be used with minor modifications 13,14. Flat bottom microtitre plates (Nunc Maxisorb, Nunc, Finland) are coated with 20 μg/ml purified capsular polysaccharide (American Type Culture Collection, Manassas, Virginia, USA) in 0.01M phosphate buffered saline (PBS), pH 7.2, for 5 hours at 37oC and then stored at 4oC. Plates are washed five times with PBS, pH7.2, with 0.05% Tween-20 after each stage. Test sera are diluted 1:50 in 1% bovine serum albumin, 0.05% Tween-20 in PBS containing 10 μg/ml C-polysaccharide (Statens Seruminstitut, Copenhagen, Denmark) and 20 μg/ml polysaccharide of serotypes 22F (American Type Culture Collection) incubated for 30 mins at room temperature. Test sera are aliquoted onto the plate in duplicate in 8 three-fold dilutions and incubated at room temperature for 1 hour. A standard reference serum (89SF, Dr Carl Frasch, FDA, USA) and a control (post-vaccination serum from an individual with good responses to all vaccine serotypes) are assayed on every plate in seven 3-fold dilutions. Bound antibody is labelled with alkaline phosphataseconjugated goat anti-human IgG in a 2 hour incubation at room temperature. Bound enzyme is visualised with p-nitrophenyl phosphate in diethanolamine substrate (Sigma) for 2 hours at room temperature and the reaction is stopped with 3M NaOH. Plates are read by an ELISA reader at a wavelength of 450 nm with a reference filter of 620nm. Results are analysed by a 4-parameter logistic-log curve fit program (ELISA v1.11, Centers for Disease Control and Prevention, Atlanta, GA) and expressed in relation to the known concentrations of the reference serum.

   ELISA FOR ANTI-PSAA: The method of Tharpe et al. will be used on pairs or triplicates of sera. Flat bottom microtitre plates (Immunlon II HB, Dynatech Corp, Chantilly, VA) are coated with 2.5 μg/ml purified PsaA in 0.01M phosphate buffered saline (PBS), pH 7.2, for 16 hours at 4oC. PsaA is produced by recombination and expression in Escherichia coli of the gene encoding PsaA. Plates are washed four times with PBS, pH7.2, with 0.05% Tween-20 after each stage except blocking, when the plates are simply emptied. Plates are blocked for 1 hour at 37oC with 1% bovine serum albumin (EIA Grade, Sigma Chemical Co., St Louise, MO) 10mg/L in PBS. Test sera are diluted in 1% bovine serum albumin, 0.05% Tween-20 in PBS and incubated for 1 hour at 37oC. Test sera are assayed in duplicate in 8 two-fold dilutions and all sera from one patient are assayed on the same plate. A reference serum of high anti-PsaA concentration and a control (Sandoglobulin, Sandoz, Switzerland) are assayed on every plate in seven 2-fold dilutions. Bound antibody is labelled with mouse monoclonal anti-human IgG-Fc conjugated to horseradish peroxidase (clone PH6043, Hybridoma Reagent laboratories, Baltimore, MD) in a 2 hour incubation at 37oC. Bound enzyme is visualised with tetramethlybenzidine (TMB 1-component microwell peroxidase substrate, Kirkegaard and Perry Laboratories Inc, Gaithersburg, MD) for 30 minutes at room temperature and the reaction is stopped with 0.18M Sulphuric Acid. Plates are read by an ELISA reader at a wavelength of 450 nm with a reference filter of 620nm. Results are analysed by a 4-parameter logistic-log curve fit program (ELISA v1.11, Centers for Disease Control and Prevention, Atlanta, GA) and expressed in ELISA units as a percentage of the concentration of the reference serum.
5. Data storage Recruitment and follow-up forms will be stored in a locked study office. Information from the forms will be entered into a computer using Filemaker Pro 5.5 and will be linked on study number and visit with the laboratory data.

ELIGIBILITY:
Pilot study (study 1)

Inclusion Criteria:

A convenience sample of 40 children aged 24-36 248 months was selected from among healthy siblings of patients admitted to the 249 paediatric ward in Kilifi District Hospital and who lived within 30km of the hospital.

Exclusion Criteria:

Subjects were excluded if they had any of the following:

1. a history of invasive pneumococcal infection including pneumonia, bacteremia, or meningitis documented at the hospital;
2. a history of previous vaccination with any pneumococcal vaccine;
3. receipt of any other vaccine in the last 2 months;
4. admission to hospital in the last 3months;
5. malnutrition, as defined by a weight-for-age z-score of <-3.0; or
6. HIV infection.

Study 2

Inclusion Criteria:

Thirty children who had recovered from an episode of invasive pneumococcal disease (the Prior IPD group) were compared with 30 healthy age-matched children who had not had IPD (the Healthy Control group). Controls were selected at random from a cohort study investigating environmental and genetic susceptibility to invasive pneumococcal disease in Kilifi District Hospital. An episode of IPD was defined as admission to hospital with cultures of blood, cerebrospinal fluid (CSF) or pleural aspirate that grew S. pneumoniae.

Exclusion Criteria:

Same as for Study 1 (pilot) except that for the Prior IPD group, history of invasive pneumococcal disease was an inclusion criterion.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2004-11-04 (Actual); Primary Completion 2006-07-03 (Actual); Study Completion 2006-07-03 (Actual)

PRIMARY OUTCOMES:
Study 1 - Pilot study: Time to reach the "response threshold" in IgG concentration to serotypes 1, 6B, 14, 19F and 23F | day 0, 5, 7, 9, 11, 14 and 28 days after vaccination
  Individual response curves for each subject and each antigen will be drawn and the pre-vaccination and the maximum concentrations will be defined. The outcome variable "response threshold" is defined as the time in days to make at least one half of the total IgG response. (The total IgG response is the difference between the maximum observed antibody concentration and the starting concentration). This is a single outcome measure derived as a composite from the different antibody concentrations across the span of the study.
Study 2 Proportional IgG Response to serotypes 1, 6B, 14, 19F and 23F within 7 days | day 0, day 7, day 11 after vaccination
  The proportion of the maximal antibody response (on day 11) that has taken place by day 7 will be estimated as follows: proportional rise = C7-C0/C11-C0, where C0, C7 and C11 represent concentrations on day 0, 7 and 11 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Scott, MD, PhD, Principal Investigator — KEMRI-Wellcome Trust Collaborative Research Program
Locations (1):
- Kilifi District Hospital, Kilifi, Coast, Kenya

IPD SHARING:
Plan to Share IPD: No